CLINICAL TRIAL: NCT01290367
Title: A Prospective, Double Blind, Controlled Study Evaluating Safety and Preliminary Efficacy of a Single Injection of Adult Mesenchymal Precursor Cells (MPCs) Combined With Hyaluronan in Subjects With Chronic Discogenic Lumbar Back Pain
Brief Title: Safety and Preliminary Efficacy Study of Mesenchymal Precursor Cells (MPCs) in Subjects With Lumbar Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mesoblast, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSB-DR001
Record Dates: First submitted 2011-02-03; First posted 2011-02-07 (Estimated); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Degenerative Disc Disease
Keywords: Chronic Lumbar Back Pain; Low back pain; Back pain; Degenerative Disc Disease; Injection of Degenerated Lumbar Disc; Stem Cells; Adult Stem Cells; Allogeneic Mesenchymal Precursor cells (MPCs); Mesoblast
MeSH Terms: conditions — Intervertebral Disc Degeneration; Low Back Pain; Back Pain | interventions — Sodium Chloride; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- High Dose MPCs (Experimental): Injection of High Dose MPCs with Hyaluronic Acid
  Interventions: Biological: Single Dose MPCs Injection
- Low Dose MPCs (Experimental): Injection of Low Dose MPCs with Hyaluronic Acid
  Interventions: Biological: Single Dose MPCs Injection
- Saline injection (Sham Comparator): Injection of saline solution.
  Interventions: Procedure: Single injection of saline solution
- Hyaluronic acid injection (Placebo Comparator): Injection of hyaluronic acid solution
  Interventions: Procedure: Single injection of hyaluronic acid

INTERVENTIONS:
Biological: Single Dose MPCs Injection — Injection of Low Dose MPCs with Hyaluronic Acid into the degenerated lumbar disc's nucleus pulposus.
  Other Names: Direct MPCs Lumbar Disc Injection.; Stem Cells
  Arms: High Dose MPCs; Low Dose MPCs
Procedure: Single injection of saline solution — Intradiscal control injection with saline solution
  Other Names: Saline injection; Sham control
  Arms: Saline injection
Procedure: Single injection of hyaluronic acid — Intradiscal control injection with hyaluronic acid
  Other Names: Hyaluronic acid injection; Vehicle control
  Arms: Hyaluronic acid injection
Biological: Single Dose MPCs Injection — Injection of HighDose MPCs with Hyaluronic Acid into the degenerated lumbar disc's nucleus pulposus.
  Other Names: Stem Cells
  Arms: High Dose MPCs; Low Dose MPCs

SUMMARY:
The purpose of this study is to compare two doses of immunoselected, culture-expanded, nucleated, allogeneic adult MPCs when combined with hyaluronic acid to two control intradiscal injections in subjects with chronic low back pain due to moderate Degenerative Disc Disease (DDD) at one lumbar level from L1 to S1.

All investigational subjects in this study will undergo injection of either 6 million (M) or 18M cells in a hyaluronic acid carrier into the degenerated lumbar disc's nucleus pulposus. All control subjects will undergo an intradiscal control injection with either saline or hyaluronic acid only

DETAILED DESCRIPTION:
This is a prospective, multicenter, double blinded, controlled clinical study comparing two doses of immunoselected, culture-expanded, nucleated, allogeneic adult MPCs when combined with hyaluronic acid to two control intradiscal injections in subjects with chronic low back pain (> 6 months) due to moderate DDD at one lumbar level from L1 to S1 and unresponsive to conservative therapy for at least 3 months (including physical therapy).

After the screening and injection visits, each subject will be evaluated clinically and radiographically at 30 days, and again at 3, 6, 12, 24 and 36 months after injection.

Subjects will be evaluated at the same time points for safety.

ELIGIBILITY:
Inclusion Criteria:

1. Male or females at least 18 years of age.
2. Have the ability to understand the requirements of the study, to provide written informed consent, and to comply with the study protocol.
3. Have the ability to understand and provide written authorization for the use and disclosure of personal health information (PHI) [per Health Insurance Portability and Accountability Act (HIPAA) privacy ruling in the US].
4. Have chronic low back pain for at least 6 months.
5. Have documented symptomatic diagnosis of DDD of one level from L1-S1 as determined by a change in disc hydration on MRI compared to normal disc with or without an annular fissure or a contained disc herniation.
6. Have failed 3 months of non-operative low back pain management.
7. Disc height loss of <30% compared to a normal adjacent disc based upon radiographic evaluation.
8. Pre-treatment baseline low back pain of at least 40 mm on a 100 mm visual analog scale.
9. Low back pain greater than leg pain.
10. Pre-treatment baseline Oswestry Disability Index Questionnaire score of at least 30 on the 100-point questionnaire.

Exclusion Criteria:

1. Female subjects who are pregnant or nursing, or women planning to become pregnant during the first year (12 months) following surgery.
2. Have a current or prior history within the last 3 years of neoplasm (excluding basal cell carcinoma) and/or any active neoplasm within the last 24 months, prior to screening.
3. Patients with compressive pathology due to stenosis or frankly herniated disc or sequestered discs are not candidates.
4. Intact disc bulge/protrusion or focal herniation at the symptomatic level (s) > 3 mm or presence of disc extrusion or sequestration.
5. Lumbar spondylitis or other undifferentiated spondyloarthropathy.
6. Have undergone a previous surgery at the involved levels.
7. Any lumbar intradiscal injection procedure (e.g., injection of corticosteroids, methylene blue, dextrose, or glucosamine and chondroitin sulfate). Discography may be performed, but must be done at least 2 weeks or more prior to the MPC injection procedure.
8. Have an acute fracture of the spine at the time of enrollment in the study.
9. Have a history of epidural steroid injections within 1 week prior to study treatment.
10. Have a known history of hypersensitivity or anaphylactic reaction to murine or bovine products or dimethyl sulfoxide (DMSO).
11. Have a positive screen for human immunodeficiency virus (HIV) antibodies.
12. Have a known history of hypersensitivity or anaphylactic reaction to Hyaluronan.
13. Have a current or prior history within the last 3 years of neoplasm (excluding basal cell carcinoma) and/or any active neoplasm within the last 24 months, prior to screening.
14. Have been a recipient of prior stem cell/progenitor cell therapy or other biological intervention to repair the target intervertebral disc.
15. Are transient or has been treated in the last 6 months before enrollment for alcohol and/or drug abuse in an inpatient substance abuse program.
16. Currently incarcerated (prisoners).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-08; Primary Completion 2013-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
To determine the overall safety of MPCs plus carrier using physical examinations, vital signs, treatment emergent adverse events (TEAEs), and the results of clinical lab tests (hematology, serum chemistry, inflammation, and immunology). | 3 years

SECONDARY OUTCOMES:
To evaluate the change of treated lumbar intervertebral discs using Magnetic Resonance Imaging (MRI) at 6 months post injection of MPCs. | 6 - 36 Months
To evaluate the effectiveness of MPCs in reducing chronic lumbar back pain using the visual analog scale (VAS). | 1 - 36 Months

CONTACTS AND LOCATIONS:
Overall Officials: Roger Brown, Study Director — Mesoblast, Ltd.
Locations (14):
- United States (13):
  - Arizona Pain Specialists, Scottsdale, Arizona
  - UC Davis Spine Center, Sacramento, California
  - The Spine Institute, Santa Monica, California
  - IPM Medical Group, Inc., Walnut Creek, California
  - Denver Spine, Denver, Colorado
  - Rocky Mountain Associates in Orthopedic Medicine, P.C., Loveland, Colorado
  - Emory University School of Medicine, Atlanta, Georgia
  - Carolina Neurosurgery and Spine Associates, Charlotte, North Carolina
  - Central Texas Spine Institute, Austin, Texas
  - Richmond Bone and Joint Clinic, Memorial Hermann Medical Group, Richmond, Texas
  - Virginia Spine Research Institute, Inc., Richmond, Virginia
  - Washington Center for Pain Management, Edmonds, Washington
  - The Center for Pain Relief, Inc., Charleston, West Virginia
- Monash Medical Center, Clayton, Victoria, Australia

REFERENCES:
- See also: Sponsor Website — http://www.mesoblast.com